CLINICAL TRIAL: NCT06068023
Title: The ADAPTA Study: ADjuvant chemotherAPy After Curative Intent resecTion of Ampullary Cancer. A Pan-European Prospective Multicenter Double Single Arm Cohort Study.
Brief Title: The ADAPTA Study: ADjuvant chemotherAPy After Curative Intent resecTion of Ampullary Cancer.
Acronym: ADAPTA
Status: Recruiting | Type: Observational
Sponsor: Fondazione Poliambulanza Istituto Ospedaliero (Other)
Collaborators: Associazione Italiana per la Ricerca sul Cancro (Other)
Responsible Party: Sponsor
Other Study IDs: ADAPTA
Record Dates: First submitted 2023-08-29; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Ampullary Adenocarcinoma
Keywords: pancreatobiliary-type; intestinal-type; mixed/hybrid-type; adjuvant chemotherapy; CAPOX; FOLFIRINOX
MeSH Terms: interventions — folfirinox; Leucovorin; Fluorouracil; Irinotecan; Oxaliplatin; Capecitabine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The analysis of the molecular markers through the genetic test of tumor samples will be performed (substudy).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Intestinal-type ampullary adenocarcinoma intervention: This cohort consist of patients with intestinal-type ampullary adenocarcinoma who are able to receive adjuvant chemotherapy.
  Interventions: Drug: Capox
- Intestinal-type ampullary adenocarcinoma control: This cohort consist of patients with intestinal-type ampullary adenocarcinoma who are able to receive adjuvant chemotherapy but due to logistics or patient preference, are not willing to receive adjuvant chemotherapy.
- Pancreatobiliary/mixed-type ampullary adenocarcinoma intervention: This cohort consist of patients with Pancreatobiliary/mixed-type ampullary adenocarcinoma who are able to receive adjuvant chemotherapy.
  Interventions: Drug: Folfirinox
- Pancreatobiliary/mixed-type ampullary adenocarcinoma control: This cohort consist of patients with Pancreatobiliary/mixed-type ampullary adenocarcinoma who are able to receive adjuvant chemotherapy but due to logistics or patient preference, are not willing to receive adjuvant chemotherapy.

INTERVENTIONS:
Drug: Folfirinox — Patients meeting the criteria of post-operative adenocarcinoma of the ampulla of Vater will be enrolled, with adjuvant chemotherapy commencing within 8 weeks of recovery from surgery. Those undergoing palliative intent surgery or palliative chemotherapy are ineligible for the ADAPTA study.
  The ADAPTA study's adjuvant chemotherapy involves 8-12 FOLFIRINOX cycles (Arm 2) repeated 2 weeks. Given patient outcomes, 8 cycles of FOLFIRINOX are deemed sufficient due to completion challenges in prior research. FOLFIRINOX regimen mirrors the modified version from the ACCORD/PRODIGE trial for metastatic pancreatic cancer. This trial adapts mFOLFIRINOX for standard practice.
  Other Names: leucovorin calcium (folinic acid), fluorouracil, irinotecan hydrochloride, and oxaliplatin.
  Groups: Pancreatobiliary/mixed-type ampullary adenocarcinoma intervention
Drug: Capox — or 8 CAPOX cycles (Arm 1) every 3 weeks.
  Other Names: Capecitabine and oxaliplatin
  Groups: Intestinal-type ampullary adenocarcinoma intervention

SUMMARY:
Ampullary adenocarcinoma (AAC) is a rare gastrointestinal cancer with varying survival rates, particularly the aggressive pancreatobiliary (PB) subtype. Adjuvant therapy benefits only PB and mixed subtype patients, while prospective studies are required for validation. A study proposes tailored adjuvant treatments (CAPOX for intestinal subtype, FOLFIRINOX for PB and mixed subtypes) based on histopathology to enhance survival, also exploring molecular sub-studies for deeper insights.

DETAILED DESCRIPTION:
Background:

Ampullary adenocarcinoma(AAC) is rare. 5-year survival rates of 30% to 70% are seen after resection. This broad range of survival could be explained by the morphological heterogeneity in the three subtypes of AAC (pancreatobiliary, intestinal and mixed subtype), which complicates the prediction of individual prognosis and clinical decision making with regard to adjuvant therapy. To date there are no prospective studies to elucidate whether adjuvant chemotherapy improves survival in these patients.

Methods/design:

The ADAPTA study is a phase II prospective single arm multicenter cohort study including 200 patients with resected AAC (100 patients with intestinal subtype, and 100 with pancreatobiliary- and mixed subtype). All patients will be treated with CAPOX/ FOLFIRINOX respectively. Outcomes will be compared after propensity score matching to data of all patients in consecutive participating centers not treated according to the proposed regime.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with histologically or cytologically confirmed AAC with subtyping of pancreatobiliary/mixed subtype or intestinal subtype
* After curative resection for ampullary cancer without metastatic disease.
* WHO performance status 0 or 1
* Able and willing to receive adjuvant chemotherapy
* R0/ R1 resection
* Age ≥ 18 years
* Written informed consent

Exclusion Criteria:

* Prior radiotherapy, chemotherapy, or resection for AAC.
* Previous malignancy (excluding non-melanoma skin cancer), unless no evidence of disease and diagnosed more than 5 years before diagnosis of AAC.
* Pregnancy.
* R2 resection.
* Adjuvant chemotherapy started more than 12 weeks after surgery (aim to start within 8 weeks)
* Serious concomitant systemic disorders that would compromise the safety of the patient or his/her ability to complete the study, at the discretion of the investigator.
* Known hypersensitivity or contraindications against capecitabine, 5 FU, Irinotecan, or Oxaliplatin
* Inadequate organ functions, characterized by:

  * Leucocytes (WBC) < 3.0 X 109/l
  * Neutrophils < 1.500 (count per microliter of blood)
  * Platelets < 100 x 109 /l
  * Hemoglobin < 8 mmol/l
  * Renal function: E-GFR < 50 ml/min (serum creatinine < 1.5 x UNL)
  * cholestasis with elevated levels of bilirubin and/or alkaline phosphatase > 3x UNL (can be improved by biliary drainage if necessary)
  * elevated transaminases (ALAT/ASAT) ≥ 5 x UNL
  * hypoalbuminemia < 2.5 g/dl
  * Inadequate coagulation status INR > 2 or Quick < 50%, aPTT >50 sec in the absence of any drugs interfering with coagulation such as acenocoumarin, warfarin, phenprocoumon, NMH or UFH.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible patients are adult non-pregnant patients with a good WHO performance score and have (borderline) resectable non-metastatic ampullary cancer.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (3y) | 3 years
  Disease-free survival (DFS) refers to the length of time after treatment for a disease in months, such as cancer, during which no signs or symptoms of the disease recur or progress. It is a crucial measure in assessing the effectiveness of a treatment regimen in preventing the return of the disease. In cancer contexts, DFS focuses on the period without disease recurrence or progression, highlighting the success of the treatment in controlling the illness.

SECONDARY OUTCOMES:
Overall survival (3y) | 3 years
  Overall survival (OS) is a critical medical outcome that measures the length of time in months from the start of treatment or diagnosis until a patient's death due to any cause. It provides a comprehensive view of the effectiveness of a treatment or intervention in extending a patient's life expectancy. OS is a fundamental endpoint in clinical trials and medical research, reflecting the real-world impact of medical strategies on patients' survival outcomes.
Disease-free survival (5y) | 5 years
  Disease-free survival (DFS) refers to the length of time in months after treatment for a disease, such as cancer, during which no signs or symptoms of the disease recur or progress. It is a crucial measure in assessing the effectiveness of a treatment regimen in preventing the return of the disease. In cancer contexts, DFS focuses on the period without disease recurrence or progression, highlighting the success of the treatment in controlling the illness.
Overall survival (5y) | 5 years
  Overall survival (OS) is a critical medical outcome that measures the length of time in months from the start of treatment or diagnosis until a patient's death due to any cause. It provides a comprehensive view of the effectiveness of a treatment or intervention in extending a patient's life expectancy. OS is a fundamental endpoint in clinical trials and medical research, reflecting the real-world impact of medical strategies on patients' survival outcomes.
Quality of Life questionnaire (qualitative outcome) | 3 years
  Quality of life (QoL) is an essential outcome measure in clinical trials that assesses the overall well-being and satisfaction of patients throughout the course of a medical intervention or treatment. It encompasses various physical, emotional, social, and functional aspects of a patient's life, beyond just medical outcomes. QoL assessments provide valuable insights into how a treatment affects patients' daily functioning, emotional state, pain levels, social interactions, and overall sense of health and happiness. The questionnaires utilized in the ADAPTA study are the EQ-5D and the QLQ-C30.

CONTACTS AND LOCATIONS:
Overall Officials: Moh'd Abu Hilal, MD, PhD, Principal Investigator — Fondazione Poliambulanza Instituto Ospedaliero
Locations (1):
- Fondazione Poliambulanza, Brescia, BS, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Upon reasonable request, the corresponding author can be contacted.

REFERENCES:
- [Background] Zhou J, Hsu CC, Winter JM, Pawlik TM, Laheru D, Hughes MA, Donehower R, Wolfgang C, Akbar U, Schulick R, Cameron J, Herman JM. Adjuvant chemoradiation versus surgery alone for adenocarcinoma of the ampulla of Vater. Radiother Oncol. 2009 Aug;92(2):244-8. doi: 10.1016/j.radonc.2009.05.006. Epub 2009 Jun 21. PMID 19541379
- [Background] Neoptolemos JP, Moore MJ, Cox TF, Valle JW, Palmer DH, McDonald AC, Carter R, Tebbutt NC, Dervenis C, Smith D, Glimelius B, Charnley RM, Lacaine F, Scarfe AG, Middleton MR, Anthoney A, Ghaneh P, Halloran CM, Lerch MM, Olah A, Rawcliffe CL, Verbeke CS, Campbell F, Buchler MW; European Study Group for Pancreatic Cancer. Effect of adjuvant chemotherapy with fluorouracil plus folinic acid or gemcitabine vs observation on survival in patients with resected periampullary adenocarcinoma: the ESPAC-3 periampullary cancer randomized trial. JAMA. 2012 Jul 11;308(2):147-56. doi: 10.1001/jama.2012.7352. PMID 22782416
- [Background] Bolm L, Ohrner K, Nappo G, Ruckert F, Zimmermann C, Rau BM, Petrova E, Honselmann KC, Lapshyn H, Bausch D, Weitz J, Sandini M, Keck T, Zerbi A, Distler M, Wellner UF. Adjuvant therapy is associated with improved overall survival in patients with pancreatobiliary or mixed subtype ampullary cancer after pancreatoduodenectomy - A multicenter cohort study. Pancreatology. 2020 Apr;20(3):433-441. doi: 10.1016/j.pan.2020.01.009. Epub 2020 Jan 21. PMID 31987649
- [Background] Conroy T, Hammel P, Hebbar M, Ben Abdelghani M, Wei AC, Raoul JL, Chone L, Francois E, Artru P, Biagi JJ, Lecomte T, Assenat E, Faroux R, Ychou M, Volet J, Sauvanet A, Breysacher G, Di Fiore F, Cripps C, Kavan P, Texereau P, Bouhier-Leporrier K, Khemissa-Akouz F, Legoux JL, Juzyna B, Gourgou S, O'Callaghan CJ, Jouffroy-Zeller C, Rat P, Malka D, Castan F, Bachet JB; Canadian Cancer Trials Group and the Unicancer-GI-PRODIGE Group. FOLFIRINOX or Gemcitabine as Adjuvant Therapy for Pancreatic Cancer. N Engl J Med. 2018 Dec 20;379(25):2395-2406. doi: 10.1056/NEJMoa1809775. PMID 30575490
- [Background] Overman MJ, Varadhachary GR, Kopetz S, Adinin R, Lin E, Morris JS, Eng C, Abbruzzese JL, Wolff RA. Phase II study of capecitabine and oxaliplatin for advanced adenocarcinoma of the small bowel and ampulla of Vater. J Clin Oncol. 2009 Jun 1;27(16):2598-603. doi: 10.1200/JCO.2008.19.7145. Epub 2009 Jan 21. PMID 19164203
- [Background] Moekotte AL, Malleo G, van Roessel S, Bonds M, Halimi A, Zarantonello L, Napoli N, Dreyer SB, Wellner UF, Bolm L, Mavroeidis VK, Robinson S, Khalil K, Ferraro D, Mortimer MC, Harris S, Al-Sarireh B, Fusai GK, Roberts KJ, Fontana M, White SA, Soonawalla Z, Jamieson NB, Boggi U, Alseidi A, Shablak A, Wilmink JW, Primrose JN, Salvia R, Bassi C, Besselink MG, Abu Hilal M. Gemcitabine-based adjuvant chemotherapy in subtypes of ampullary adenocarcinoma: international propensity score-matched cohort study. Br J Surg. 2020 Aug;107(9):1171-1182. doi: 10.1002/bjs.11555. Epub 2020 Apr 7. PMID 32259295
- See also: ADAPTA website — https://isgaca.com/adapta/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-17): https://cdn.clinicaltrials.gov/large-docs/23/NCT06068023/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-17): https://cdn.clinicaltrials.gov/large-docs/23/NCT06068023/ICF_001.pdf